CLINICAL TRIAL: NCT00001224
Title: Immunologic Analysis of Intra-Ocular Tissue
Brief Title: Analysis of Eye Tissue
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 870104; 87-EI-0104
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-09

CONDITIONS: Eye Disease; Inflammation; Uveitis
Keywords: Ocular Inflammatory Disease; Cataracts; Vitrectomy; Extracapsular; Cataract Surgery; Uveitis; Lenticular Opacity; Vitreal Opacity
MeSH Terms: conditions — Eye Diseases; Inflammation; Uveitis; Cataract

SUMMARY:
The purpose of this investigation is to better understand the inflammatory process that occurs in uveitis (eye inflammation) through study of eye tissues.

Patients with uveitis sometimes develop cataracts (clouding of the lens of the eye) or clouding of the vitreous-the gel-like material behind the lens-that can impair eyesight. Those who require cataract surgery or vitrectomy are eligible for this study. Samples of eye tissue and fluid normally removed during standard surgical procedures for these conditions will be given to researchers instead of discarded, as is usually done.

Before surgery, patients will undergo routine preoperative tests, including chest X-ray, electrocardiogram, blood tests and urinalysis. They will also have an eye examination and photographs taken of the retina. Other tests that may be performed include fluorescein angiography to evaluate the blood vessels of the retina; ultrasound to examine the back of the eye; and a gallium scan to evaluate inflammation.

Immune cells in the blood and eye tissue will be compared and categorized by disease. The eye fluid will be examined for substances involved in the inflammatory process. These studies may provide information that will lead to improved methods of diagnosis and treatment.

DETAILED DESCRIPTION:
The purpose of this project is to evaluate intra-ocular tissue such as iris or vitreous from uveitis patients in order to analyze the type and character of the inflammatory response. Patients with a history of uveitis who require cataract surgery or vitreous surgery because of the clinical complications of inflammation, will be entered in this study. The lymphocyte subsets in the peripheral blood and ocular tissue will be compared and categorized by disease. The presence of soluble lymphokines in the intra-ocular fluid will be analyzed. Long term cell cultures of vitreal cells will be attempted to define the T-cell receptors. In addition, a portion of iris tissue or vitreous cells will be frozen to establish a tissue library of uveitis.

ELIGIBILITY:
Patients of either sex will be admitted to this study.

All patients should have a previous history of uveitis.

The patient must have lenticular or vitreal opacities which are significantly impairing their vision and for which surgical removal of the opacity has a reasonable chance of improving the vision.

Patients should have vision of 20/80 or worse.

Patients may have any of the following syndromes: anterior uveitis, including HLA-B27-associated iritis and juvenile rheumatoid arthritis, ocular sarcoid, intermediate uveitis and pars planitis, birdshot retinochoroidopathy, Behcet's disease, Vogt-Koyanagi-Harada's syndrome, sympathic ophthalmia and idiopathic posterior uveitis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Start 1987-07; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Chan CC, Nussenblatt RB, Fujikawa LS, Palestine AG, Stevens G Jr, Parver LM, Luckenbach MW, Kuwabara T. Sympathetic ophthalmia. Immunopathological findings. Ophthalmology. 1986 May;93(5):690-5. doi: 10.1016/s0161-6420(86)33694-7. PMID 3523359
- [Background] Whitcup SM, Stark-Vancs V, Wittes RE, Solomon D, Podgor MJ, Nussenblatt RB, Chan CC. Association of interleukin 10 in the vitreous and cerebrospinal fluid and primary central nervous system lymphoma. Arch Ophthalmol. 1997 Sep;115(9):1157-60. doi: 10.1001/archopht.1997.01100160327010. PMID 9298057
- [Background] George RK, Chan CC, Whitcup SM, Nussenblatt RB. Ocular immunopathology of Behcet's disease. Surv Ophthalmol. 1997 Sep-Oct;42(2):157-62. doi: 10.1016/s0039-6257(97)00026-x. PMID 9381369